CLINICAL TRIAL: NCT00149864
Title: Multicenter, Open-label Follow-up Study on the Safety of Enteric-coated Mycophenolate Sodium in Maintenance Renal Transplant Patients
Brief Title: Follow-up Study of Safety of Enteric-coated Mycophenolate Sodium in Patients Who Successfully Completed Study CERL080A302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A302E
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Renal Transplant
Keywords: Renal Transplant, adults, immunosuppressant
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolate sodium (enteric coated)

SUMMARY:
Aim of study is to collect long term safety data on enteric-coated mycophenolate sodium 720 mg bid in combination with cyclosporine with/without steroids in regard to adverse events, serious adverse events, and patient and graft survival. After successful completion of the study CERL080A302, patients who previously were receiving enteric-coated mycophenolate sodium or MMF were given opportunity to remain on enteric-coated mycophenolate sodium or convert MMF to enteric-coated mycophenolate sodium.

ELIGIBILITY:
Inclusion Criteria:

-First cadaveric, living unrelated or living related donor kidney transplant recipients who completed study CERL080A302

Exclusion Criteria:

* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2000-02; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To assess the incidence and severity of GI adverse events (AEs) and neutropenia in the first 3 months of treatment in maintenance renal transplant patients.

SECONDARY OUTCOMES:
Safety/efficacy based on adverse event (AE) reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis